CLINICAL TRIAL: NCT02409290
Title: STREAM: The Evaluation of a Standard Treatment Regimen of Anti-tuberculosis Drugs for Patients With MDR-TB
Brief Title: The Evaluation of a Standard Treatment Regimen of Anti-tuberculosis Drugs for Patients With MDR-TB
Acronym: STREAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IUATLD, Inc (Other)
Collaborators: Medical Research Council (Other Government); Institute of Tropical Medicine, Belgium (Other); Liverpool School of Tropical Medicine (Other); Rede TB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78372190/18148631 (Stage 1/2)
Record Dates: First submitted 2015-03-31; First posted 2015-04-06 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: MDR-TB
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Moxifloxacin; Clofazimine; Ethambutol; Pyrazinamide; Isoniazid; Prothionamide; Kanamycin; Levofloxacin; bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen A (Active Comparator): Regimen A locally-used WHO-approved MDR-TB regimen in accordance with 2011 WHO MDR-TB treatment guidelines.
  Interventions: Drug: Regimen A locally-used WHO-approved MDR-TB regimen (2011 guideline)
- Regimen B (Active Comparator): Regimen B is based on the regimen described by Van Deun 2010. With Version 8.0 of the protocol Regimen B (Regimen Bmox) is modified by replacement of moxifloxacin with levofloxacin (Regimen Blev). Regimen B without specification of which fluoroquinolone is in the regimen refers to either (Bmox or Blev).
  Product and dose for [<33 kg, 33-50kg, >50 kg] respectively:
  Moxifloxacin [400mg, 600mg, 800mg] OR Levofloxacin [750mg, 750mg,1000mg]; Clofazimine [50mg,100mg,100mg]; Ethambutol [800mg,800mg,1200mg]; Pyrazinamide [1000mg,1500mg, 2000mg]; Isoniazid 300mg, 400mg, 600mg]; Prothionamide [250mg,500mg,750mg]; Kanamycin [15mg per kilogram body weight (maximum 1g)].
  Interventions: Drug: Moxifloxacin; Drug: Clofazimine; Drug: Ethambutol; Drug: Pyrazinamide; Drug: Isoniazid; Drug: Prothionamide; Drug: Kanamycin; Drug: Levofloxacin
- Regimen C (Experimental): Regimen C is a 40-week all-oral regimen consisting of bedaquiline, clofazimine, ethambutol, levofloxacin, and pyrazinamide given for 40 weeks supplemented by isoniazid and prothionamide for the first 16 weeks (intensive phase).
  Product and dose for [<33kg, 33-50kg, >50 kg] respectively:
  Bedaquiline 400mg once daily for first 14 days/200 mg thrice weekly thereafter; Levofloxacin [750mg, 750mg,1000mg]; Clofazimine [50mg, 100mg, 100mg]; Ethambutol [800mg, 800mg, 1200mg]; Pyrazinamide [1000mg,1500mg, 2000mg]; Isoniazid [300mg, 400mg, 600mg]; Prothionamide [250mg, 500mg,750mg].
  Interventions: Drug: Clofazimine; Drug: Ethambutol; Drug: Pyrazinamide; Drug: Isoniazid; Drug: Prothionamide; Drug: Levofloxacin; Drug: Bedaquiline
- Regimen D (Experimental): Regimen D is a 28-week regimen consisting of bedaquiline, clofazimine, levofloxacin, and pyrazinamide given for 28 weeks supplemented by isoniazid and kanamycin for the first 8 weeks (intensive phase).
  Product and dose for [<33kg, 33 to<40kg, 40-50kg, >50-60 kg, >60 kg] respectively:
  Bedaquiline 400mg once daily for first 14 days/200mg thrice weekly thereafter; Levofloxacin [750mg, 750mg, 750mg, 1000mg, 1000mg]; Clofazimine [50mg, 100mg, 100mg, 100mg, 100mg]; Pyrazinamide [1000mg,1500mg, 1500mg, 2000mg, 2000mg]; Isoniazid [400mg, 500mg, 600mg, 800mg, 900mg]; Kanamycin [15 mg per kilogram body weight (maximum 1g)].
  Interventions: Drug: Clofazimine; Drug: Pyrazinamide; Drug: Isoniazid; Drug: Kanamycin; Drug: Levofloxacin; Drug: Bedaquiline

INTERVENTIONS:
Drug: Regimen A locally-used WHO-approved MDR-TB regimen (2011 guideline) — Drug: Locally-used WHO-approved MDR-TB regimen
  Arms: Regimen A
Drug: Moxifloxacin — Moxifloxacin is an 8-methoxy quinolone, and an anti-bacterial fluoroquinolone
  Other Names: Avelox
  Arms: Regimen B
Drug: Clofazimine — Clofazimine, is an antileprosy and anti-bacterial agent. Its chemical name is 3-(p-chloroanilino)-10-(p-chlorophenyl)-2, 10-dihydro-2-isopropyliminophenazine.
  Other Names: Lamprene
  Arms: Regimen B; Regimen C; Regimen D
Drug: Ethambutol — Ethambutol is a bacteriostatic that acts against virtually all strains of Mycobacterium tuberculosis and M. bovis and is also active against other mycobacteria such as M. Kansasii.
  Other Names: Myambutol
  Arms: Regimen B; Regimen C
Drug: Pyrazinamide — Pyrazinamide is bactericidal against intracellular mycobacterium tuberculosis. It is a prodrug that is converted into its active form, pyrazinoic acid, by a mycobacterial enzyme, pyrazinamidase, as well as through hepatic metabolism.
  Other Names: Zinamide
  Arms: Regimen B; Regimen C; Regimen D
Drug: Isoniazid — Isoniazid is a bactericidal in vitro and in vivo against actively dividing tubercle bacilli. Its primary action is to inhibit the synthesis of long-chain mycolic acids, which are unique constituents of mycobacterial cell wall.
  Other Names: Nydrazid; Isotamine
  Arms: Regimen B; Regimen C; Regimen D
Drug: Prothionamide — Prothionamide has a bacteriostatic action.
  Other Names: Peteha
  Arms: Regimen B; Regimen C
Drug: Kanamycin — Kanamycin is a bactericidal antibiotic from the group of aminoglycosides.
  Other Names: Kantrex
  Arms: Regimen B; Regimen D
Drug: Levofloxacin — Levofloxacin is a synthetic antibacterial agent of the fluoroquinolone class that acts on the DNA-DNA-gyrase complex and topoisomerase IV. It is the S (-) enantiomer of the racemic active substance ofloxacin.
  Other Names: Levaquin
  Arms: Regimen B; Regimen C; Regimen D
Drug: Bedaquiline — Bedaquiline is a novel diarylquinoline antibiotic with bactericidal activity
  Other Names: SIRTURO
  Arms: Regimen C; Regimen D

SUMMARY:
Tuberculosis (TB) is a common, infectious, bacterial disease that is spread when an infected person transmits their saliva through the air by coughing or sneezing. Despite the availability and effectiveness of affordable six-month treatments for tuberculosis (TB), the worldwide control of this disease is currently being impacted by the emergence of multidrug resistant TB (MDR-TB). MDR-TB refers to TB that is resistant to at least isoniazid and rifampicin. These are the two most powerful first-line drugs used to treat pulmonary TB. MDR-TB usually develops while a person is taking TB treatment due to either inappropriate treatment or failure of patients to comply with their treatment. This strain of drug-resistant bacteria can also be spread to other people through the air. With the incident rate of MDR-TB on the rise, there is a need to investigate optimal treatment regimens using effective drugs.

DETAILED DESCRIPTION:
The STREAM study is an international, multi-centre, parallel-group, open-label, randomised, controlled trial in patients with multi-drug resistant tuberculosis (MDR-TB) including patients with rifampicin-resistant and isoniazid-sensitive TB.

Background and Rationale:

In 2011, World Health Organisation (WHO) guidelines for the treatment for MDR-TB recommended an intensive phase of treatment based on at least four drugs known to be effective and given for a minimum of 20 months; this is referred to as the WHO 2011 long regimen. Outcomes with this approach are generally poor. In the most recent WHO TB surveillance report only 50% of MDR-TB patients were successfully treated and a recent meta-analysis reported on average 62% successful outcome and a mortality of 11%.

In 2010, Van Deun et al (2010) reported excellent long-term outcomes in a cohort of over 200 patients in Bangladesh with MDR-TB who were treated with a regimen given for only nine to 11 months. Such a regimen, if successful, would represent a considerable advance over current practice. Evaluation of this regimen is the objective of Stage 1 of STREAM.

In 2016, following review of the available data, the WHO MDR TB treatment guidelines were modified to recommend a 9-12 month shortened regimen under specific conditions similar to Regimen B used in STREAM Stage 1 (referred to as the WHO 2016 short regimen).

Bedaquiline is a novel diarylquinoline antibiotic with bactericidal activity. In a phase II trial of patients with MDR-TB time to culture conversion was significantly less in patients receiving bedaquiline compared to those receiving an optimised background regimen only (Diacon et al (2012). In December 2012 the US Food and Drug Administration (FDA) approved bedaquiline as part of the treatment regimen for MDR-TB when other agents are unavailable. Stage 2 of STREAM was designed to investigate ways in which Regimen B could be improved either by removing the second-line injectable, which is associated with severe drug toxicity, or by shortening the regimen to 6 months.

Treatments that are evaluated within the STREAM trial include:

Regimen A The locally-used MDR-TB regimen in accordance with 2011 WHO MDR-TB treatment guidelines.

Regimen B is based on the regimen described by Van Deun 2010. At the start of STREAM this consisted of clofazimine, ethambutol, moxifloxacin, and pyrazinamide given for 40 weeks, supplemented by isoniazid, kanamycin, and prothionamide in the first 16 weeks (intensive phase). ); this combination is referred to as Regimen Bmox. With Version 8.0 of the protocol Regimen B is modified by replacement of moxifloxacin with levofloxacin (referred to as Regimen Blev). Regimen B without specification of which fluoroquinolone is in the regimen refers to either (Bmox or Blev).

Regimen C is a 40-week all-oral regimen consisting of bedaquiline, clofazimine, ethambutol, levofloxacin, and pyrazinamide given for 40 weeks supplemented by isoniazid and prothionamide for the first 16 weeks (intensive phase).

Regimen D is a 28-week regimen consisting of bedaquiline, clofazimine, levofloxacin, and pyrazinamide given for 28 weeks supplemented by isoniazid and kanamycin for the first 8 weeks (intensive phase).

The primary objectives of the STREAM2 trial are:

To assess whether the proportion of participants with a favourable efficacy outcome at week 76 on Regimen C is non-inferior to that on Regimen B

Study Population: Stage 2 will aim to randomise at least 200 patients to each of Regimens B and C.

All patients will be followed up to Week 132. The primary analysis will be based on the data accrued to Week 76 and is based on the proportion of patients with a favourable outcome at that time point ; the data accrued to Week 132 will be used in secondary analyses.

Although the STREAM study is an open-label study, wherever possible it will be conducted masked to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Consent: Is willing and able to give informed consent to participate in the trial treatment and follow-up (signed or witnessed consent if the patient is illiterate). If the patient is below the age of consent (according to local regulations), the parent/caregiver should be able and willing to give consent, and the patient be informed about the study and asked to give positive assent, if feasible
2. Age: Is aged 18 years or older (Stage 1) or 15 years or older (Stage 2)
3. AFB or GeneXpert results: Has a positive AFB sputum smear result at screening (at least scanty), or a positive GeneXpert result (with a cycle threshold (Ct) value of 25 or lower) from a test performed at screening or from a test performed within the four weeks prior to screening
4. Has evidence of resistance to rifampicin either by line probe assay (Hain Genotype), GeneXpert or culture-based drug susceptibility testing (DST), from a test performed at screening or from a test performed within the four weeks prior to screening
5. Is willing to have an HIV test and, if positive, is willing to be treated with ART in accordance with the national policies but excluding ART contraindicated for use with bedaquiline
6. Is willing to use effective contraception: pre-menopausal women or women whose last menstrual period was within the preceding year, who have not been sterilised must agree to use a barrier method or an intrauterine device unless their partner has had a vasectomy; men who have not had a vasectomy must agree to use condoms. In Stage 2 pre-menopausal women or women whose last menstrual period was within the preceding year, who have not been sterilised must agree to use two methods of contraception, for example a hormonal method and a barrier method
7. Resides in the area and expected to remain for the duration of the study.
8. Has had a chest X-ray that is compatible with a diagnosis of pulmonary TB (if such a chest X-ray taken within 4 weeks of randomisation is available, a repeat X-ray is not required)
9. Has normal K+, Mg2+ and corrected Ca2+ at screening.

Exclusion Criteria:

1. Is infected with a strain of M. tuberculosis resistant to second-line injectables by line probe assay (Hain Genotype) from a test performed at screening or from a test performed within the four weeks prior to screening
2. Is infected with a strain of M. tuberculosis resistant to fluoroquinolones by line probe assay (Hain Genotype) from a test performed at screening or from a test performed within the four weeks prior to screening
3. Has tuberculous meningitis or bone and joint tuberculosis
4. Is critically ill, and in the judgment of the investigator, unlikely to survive more than 4 months
5. Is known to be pregnant or breast-feeding
6. Is unable or unwilling to comply with the treatment, assessment, or follow-up schedule
7. Is unable to take oral medication
8. Has AST or ALT more than 5 times the upper limit of normal for Stage 1, and AST or ALT more than 3 times the upper limit of normal for Stage 2
9. Has any condition (social or medical) which in the opinion of the investigator would make study participation unsafe
10. In the investigator's opinion the patient is likely to be eligible for treatment with bedaquiline according to local guidelines due to a pre-existing medical condition such as hearing loss or renal impairment
11. Is taking any medications contraindicated with the medicines in any trial regimen
12. Has a known allergy to any fluoroquinolone antibiotic
13. Is currently taking part in another trial of a medicinal product
14. Has a QT or QTcF interval at screening or immediately prior to randomisation of more than or equal to 500 ms for Stage 1, and more than or equal to 450 ms for Stage 2

    In addition to the criteria above, for Stage 2 only, a patient will not be eligible for randomisation to the study if he/she:
15. Has experienced one or more of the following risk factors for QT prolongation:

    * A confirmed prolongation of the QT or QTcF more than or equal to 450 ms in the screening ECG (retesting to reassess eligibility will be allowed once using an unscheduled visit during the screening phase)
    * Pathological Q-waves (defined as Q-wave more than 40 ms or depth more than 0.4-0.5 mV)
    * Evidence of ventricular pre-excitation (e.g., Wolff Parkinson White syndrome)
    * Electrocardiographic evidence of complete or clinically significant incomplete left bundle branch block or right bundle branch block
    * Evidence of second or third degree heart block
    * Intraventricular conduction delay with QRS duration more than 120 ms
    * Bradycardia as defined by sinus rate less than 50 bpm
    * Personal or family history of Long QT Syndrome
    * Personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, with the exception of sinus arrhythmia
    * Syncope (i.e. cardiac syncope not including syncope due to vasovagal or epileptic causes)
    * Risk factors for Torsades de Pointes (e.g., heart failure, hypokalaemia, or hypomagnesemia)
16. Has received treatment for MDR-TB in the 12 weeks prior to screening, other than the maximum permitted treatment specified in Section 5.2.1
17. Has a history of cirrhosis and classified as Child's B or C at screening or a bilirubin more than 1.5 times upper limit of normal.
18. Has an estimated creatinine clearance (CrCl) less than 30 mL/min based on the Cockcroft-Gault equation
19. Is HIV positive and has a CD4 count less than 50 cells/mm3
20. Has pancreatic amylase elevation more than two times above the upper limit of normal
21. Has a history of alcohol and/or drug abuse
22. Has had previous treatment with bedaquiline
23. Has taken rifampicin in the seven days prior to randomisation
24. There has been a delay of more than four weeks between the screening consent and randomisation
25. Is an employee or family member of the investigator or study site staff with direct involvement in the proposed study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Meredith, MD, Principal Investigator — Medical Research Council; Andrew Nunn, PhD, Principal Investigator — Medical Research Council
Locations (13):
- Ethiopia (2):
  - Armauer Hanssen Research Institute, Addis Ababa
  - St. Peter's Tuberculosis Specializes Hospital, Addis Ababa
- JSC National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- India (3):
  - BJ Medical College Civil Hospital, Ahmedabad
  - The National Institute for Research in Tuberculosis, Chennai
  - Rajan Babu Institute for Pulmonary Medicine and Tuberculosis, New Delhi
- Institute of Phthisiopneumology 'Chiril Draganiuc', Chisinau, Moldova
- National Centre for Communicable Diseases, Ulaanbaatar, Mongolia
- South Africa (4):
  - King Dinizulu Hospital, Durban
  - Helen Joseph Hospital, Johannesburg
  - Doris Goodwin Hospital, Pietermaritzburg
  - Empilweni TB Hospital, Port Elizabeth
- Makerere University (Mulago Referral Hospital), Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including individual participant data and a data dictionary defining each field in the set, will be made available no later than 12 months after the end of the trial through the TBPACT data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From May 2024 at the latest.
Access Criteria: Application to CPATH as described on the website.
URL: https://c-path.org/programs/tb-pacts/

REFERENCES:
- [Background] Van Deun A, Maug AK, Salim MA, Das PK, Sarker MR, Daru P, Rieder HL. Short, highly effective, and inexpensive standardized treatment of multidrug-resistant tuberculosis. Am J Respir Crit Care Med. 2010 Sep 1;182(5):684-92. doi: 10.1164/rccm.201001-0077OC. Epub 2010 May 4. PMID 20442432
- [Background] Laserson KF, Wells CD. Reaching the targets for tuberculosis control: the impact of HIV. Bull World Health Organ. 2007 May;85(5):377-81; discussion 382-6. doi: 10.2471/blt.06.035329. PMID 17639223
- [Background] Zignol M, Hosseini MS, Wright A, Weezenbeek CL, Nunn P, Watt CJ, Williams BG, Dye C. Global incidence of multidrug-resistant tuberculosis. J Infect Dis. 2006 Aug 15;194(4):479-85. doi: 10.1086/505877. Epub 2006 Jul 12. PMID 16845631
- [Background] Wells CD, Cegielski JP, Nelson LJ, Laserson KF, Holtz TH, Finlay A, Castro KG, Weyer K. HIV infection and multidrug-resistant tuberculosis: the perfect storm. J Infect Dis. 2007 Aug 15;196 Suppl 1:S86-107. doi: 10.1086/518665. PMID 17624830
- [Background] Guidelines for the Programmatic Management of Drug-Resistant Tuberculosis: 2011 Update. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK148644/ PMID 23844450
- [Background] Seung KJ, Omatayo DB, Keshavjee S, Furin JJ, Farmer PE, Satti H. Early outcomes of MDR-TB treatment in a high HIV-prevalence setting in Southern Africa. PLoS One. 2009 Sep 25;4(9):e7186. doi: 10.1371/journal.pone.0007186. PMID 19779624
- [Background] Chiang CY, Enarson DA, Yu MC, Bai KJ, Huang RM, Hsu CJ, Suo J, Lin TP. Outcome of pulmonary multidrug-resistant tuberculosis: a 6-yr follow-up study. Eur Respir J. 2006 Nov;28(5):980-5. doi: 10.1183/09031936.06.00125705. Epub 2006 Jul 12. PMID 16837502
- [Background] Mitnick C, Bayona J, Palacios E, Shin S, Furin J, Alcantara F, Sanchez E, Sarria M, Becerra M, Fawzi MC, Kapiga S, Neuberg D, Maguire JH, Kim JY, Farmer P. Community-based therapy for multidrug-resistant tuberculosis in Lima, Peru. N Engl J Med. 2003 Jan 9;348(2):119-28. doi: 10.1056/NEJMoa022928. PMID 12519922
- [Background] Leimane V, Riekstina V, Holtz TH, Zarovska E, Skripconoka V, Thorpe LE, Laserson KF, Wells CD. Clinical outcome of individualised treatment of multidrug-resistant tuberculosis in Latvia: a retrospective cohort study. Lancet. 2005 Jan 22-28;365(9456):318-26. doi: 10.1016/S0140-6736(05)17786-1. PMID 15664227
- [Background] Orenstein EW, Basu S, Shah NS, Andrews JR, Friedland GH, Moll AP, Gandhi NR, Galvani AP. Treatment outcomes among patients with multidrug-resistant tuberculosis: systematic review and meta-analysis. Lancet Infect Dis. 2009 Mar;9(3):153-61. doi: 10.1016/S1473-3099(09)70041-6. PMID 19246019
- [Background] Diacon AH, Donald PR, Pym A, Grobusch M, Patientia RF, Mahanyele R, Bantubani N, Narasimooloo R, De Marez T, van Heeswijk R, Lounis N, Meyvisch P, Andries K, McNeeley DF. Randomized pilot trial of eight weeks of bedaquiline (TMC207) treatment for multidrug-resistant tuberculosis: long-term outcome, tolerability, and effect on emergence of drug resistance. Antimicrob Agents Chemother. 2012 Jun;56(6):3271-6. doi: 10.1128/AAC.06126-11. Epub 2012 Mar 5. PMID 22391540
- [Background] Mann G, Squire SB, Bissell K, Eliseev P, Du Toit E, Hesseling A, Nicol M, Detjen A, Kritski A. Beyond accuracy: creating a comprehensive evidence base for TB diagnostic tools. Int J Tuberc Lung Dis. 2010 Dec;14(12):1518-24. PMID 21144235
- [Background] Johnson JL, Hadad DJ, Boom WH, Daley CL, Peloquin CA, Eisenach KD, Jankus DD, Debanne SM, Charlebois ED, Maciel E, Palaci M, Dietze R. Early and extended early bactericidal activity of levofloxacin, gatifloxacin and moxifloxacin in pulmonary tuberculosis. Int J Tuberc Lung Dis. 2006 Jun;10(6):605-12. PMID 16776446
- [Background] Lancioni GE, Coninx F, Smeets PM. A classical conditioning procedure for the hearing assessment of multiply handicapped persons. J Speech Hear Disord. 1989 Feb;54(1):88-93. doi: 10.1044/jshd.5401.88. PMID 2521683
- [Background] Cegielski JP, Dalton T, Yagui M, Wattanaamornkiet W, Volchenkov GV, Via LE, Van Der Walt M, Tupasi T, Smith SE, Odendaal R, Leimane V, Kvasnovsky C, Kuznetsova T, Kurbatova E, Kummik T, Kuksa L, Kliiman K, Kiryanova EV, Kim H, Kim CK, Kazennyy BY, Jou R, Huang WL, Ershova J, Erokhin VV, Diem L, Contreras C, Cho SN, Chernousova LN, Chen MP, Caoili JC, Bayona J, Akksilp S; Global Preserving Effective TB Treatment Study (PETTS) Investigators. Extensive drug resistance acquired during treatment of multidrug-resistant tuberculosis. Clin Infect Dis. 2014 Oct 15;59(8):1049-63. doi: 10.1093/cid/ciu572. Epub 2014 Jul 23. PMID 25057101
- [Background] Fox GJ, Menzies D. A Review of the Evidence for Using Bedaquiline (TMC207) to Treat Multi-Drug Resistant Tuberculosis. Infect Dis Ther. 2013 Dec;2(2):123-44. doi: 10.1007/s40121-013-0009-3. Epub 2013 Aug 2. PMID 25134476
- [Background] McClure N, Dornal JC. Early identification of placenta praevia. Br J Obstet Gynaecol. 1990 Oct;97(10):959-61. doi: 10.1111/j.1471-0528.1990.tb02457.x. No abstract available. PMID 2223692
- [Background] Hillemann D, Rusch-Gerdes S, Richter E. Feasibility of the GenoType MTBDRsl assay for fluoroquinolone, amikacin-capreomycin, and ethambutol resistance testing of Mycobacterium tuberculosis strains and clinical specimens. J Clin Microbiol. 2009 Jun;47(6):1767-72. doi: 10.1128/JCM.00081-09. Epub 2009 Apr 22. PMID 19386845
- [Background] Mohamed K, Embleton A, Cuffe RL. Adjusting for covariates in non-inferiority studies with margins defined as risk differences. Pharm Stat. 2011 Sep-Oct;10(5):461-6. doi: 10.1002/pst.520. PMID 21956950
- [Background] Gumbo T, Louie A, Deziel MR, Parsons LM, Salfinger M, Drusano GL. Selection of a moxifloxacin dose that suppresses drug resistance in Mycobacterium tuberculosis, by use of an in vitro pharmacodynamic infection model and mathematical modeling. J Infect Dis. 2004 Nov 1;190(9):1642-51. doi: 10.1086/424849. Epub 2004 Sep 24. PMID 15478070
- [Background] Falagas ME, Rafailidis PI, Rosmarakis ES. Arrhythmias associated with fluoroquinolone therapy. Int J Antimicrob Agents. 2007 Apr;29(4):374-9. doi: 10.1016/j.ijantimicag.2006.11.011. Epub 2007 Jan 22. PMID 17241772
- [Background] Altin T, Ozcan O, Turhan S, Ongun Ozdemir A, Akyurek O, Karaoguz R, Guldal M. Torsade de pointes associated with moxifloxacin: a rare but potentially fatal adverse event. Can J Cardiol. 2007 Sep;23(11):907-8. doi: 10.1016/s0828-282x(07)70850-4. PMID 17876386
- [Background] Haddad PM, Anderson IM. Antipsychotic-related QTc prolongation, torsade de pointes and sudden death. Drugs. 2002;62(11):1649-71. doi: 10.2165/00003495-200262110-00006. PMID 12109926
- [Background] Florian JA, Tornoe CW, Brundage R, Parekh A, Garnett CE. Population pharmacokinetic and concentration--QTc models for moxifloxacin: pooled analysis of 20 thorough QT studies. J Clin Pharmacol. 2011 Aug;51(8):1152-62. doi: 10.1177/0091270010381498. Epub 2011 Jan 12. PMID 21228407
- [Background] Tsikouris JP, Peeters MJ, Cox CD, Meyerrose GE, Seifert CF. Effects of three fluoroquinolones on QT analysis after standard treatment courses. Ann Noninvasive Electrocardiol. 2006 Jan;11(1):52-6. doi: 10.1111/j.1542-474X.2006.00082.x. PMID 16472283
- [Background] Sherazi S, DiSalle M, Daubert JP, Shah AH. Moxifloxacin-induced torsades de pointes. Cardiol J. 2008;15(1):71-3. PMID 18651388
- [Background] Dale KM, Lertsburapa K, Kluger J, White CM. Moxifloxacin and torsade de pointes. Ann Pharmacother. 2007 Feb;41(2):336-40. doi: 10.1345/aph.1H474. Epub 2007 Feb 6. PMID 17284508
- [Background] Rubinstein E, Camm J. Cardiotoxicity of fluoroquinolones. J Antimicrob Chemother. 2002 Apr;49(4):593-6. doi: 10.1093/jac/49.4.593. No abstract available. PMID 11909831
- [Background] Morganroth J, Dimarco JP, Anzueto A, Niederman MS, Choudhri S; CAPRIE Study Group. A randomized trial comparing the cardiac rhythm safety of moxifloxacin vs levofloxacin in elderly patients hospitalized with community-acquired pneumonia. Chest. 2005 Nov;128(5):3398-406. doi: 10.1378/chest.128.5.3398. PMID 16304291
- [Background] Demolis JL, Kubitza D, Tenneze L, Funck-Brentano C. Effect of a single oral dose of moxifloxacin (400 mg and 800 mg) on ventricular repolarization in healthy subjects. Clin Pharmacol Ther. 2000 Dec;68(6):658-66. doi: 10.1067/mcp.2000.111482. PMID 11180026
- [Background] Noel GJ, Natarajan J, Chien S, Hunt TL, Goodman DB, Abels R. Effects of three fluoroquinolones on QT interval in healthy adults after single doses. Clin Pharmacol Ther. 2003 Apr;73(4):292-303. doi: 10.1016/s0009-9236(03)00009-2. PMID 12709719
- [Background] Sacco F, Spezzaferro M, Amitrano M, Grossi L, Manzoli L, Marzio L. Efficacy of four different moxifloxacin-based triple therapies for first-line H. pylori treatment. Dig Liver Dis. 2010 Feb;42(2):110-4. doi: 10.1016/j.dld.2009.05.013. Epub 2009 Oct 28. PMID 19846355
- [Background] Stass H, Dalhoff A, Kubitza D, Schuhly U. Pharmacokinetics, safety, and tolerability of ascending single doses of moxifloxacin, a new 8-methoxy quinolone, administered to healthy subjects. Antimicrob Agents Chemother. 1998 Aug;42(8):2060-5. doi: 10.1128/AAC.42.8.2060. PMID 9687407
- [Background] Alffenaar JW, de Vries PM, Luijckx GJ, van Soolingen D, van der Werf TS, van Altena R. Plasma and cerebrospinal fluid pharmacokinetics of moxifloxacin in a patient with tuberculous meningitis. Antimicrob Agents Chemother. 2008 Jun;52(6):2293-5. doi: 10.1128/AAC.01637-07. Epub 2008 Mar 24. No abstract available. PMID 18362186
- [Background] Soliman EZ, Lundgren JD, Roediger MP, Duprez DA, Temesgen Z, Bickel M, Shlay JC, Somboonwit C, Reiss P, Stein JH, Neaton JD; INSIGHT SMART Study Group. Boosted protease inhibitors and the electrocardiographic measures of QT and PR durations. AIDS. 2011 Jan 28;25(3):367-77. doi: 10.1097/QAD.0b013e328341dcc0. PMID 21150558
- [Derived] Hughes G, Young WJ, Bern H, Crook A, Lambiase PD, Goodall RL, Nunn AJ, Meredith SK. T-wave morphology abnormalities in the STREAM stage 1 trial. Expert Opin Drug Saf. 2024 Apr;23(4):469-476. doi: 10.1080/14740338.2024.2322116. Epub 2024 Mar 10. PMID 38462751
- [Derived] Nunn AJ, Phillips PPJ, Meredith SK, Chiang CY, Conradie F, Dalai D, van Deun A, Dat PT, Lan N, Master I, Mebrahtu T, Meressa D, Moodliar R, Ngubane N, Sanders K, Squire SB, Torrea G, Tsogt B, Rusen ID; STREAM Study Collaborators. A Trial of a Shorter Regimen for Rifampin-Resistant Tuberculosis. N Engl J Med. 2019 Mar 28;380(13):1201-1213. doi: 10.1056/NEJMoa1811867. Epub 2019 Mar 13. PMID 30865791
- [Derived] Moodley R, Godec TR; STREAM Trial Team. Short-course treatment for multidrug-resistant tuberculosis: the STREAM trials. Eur Respir Rev. 2016 Mar;25(139):29-35. doi: 10.1183/16000617.0080-2015. PMID 26929418
- See also: Medical Research Council at UCL's web page containing information on the trial — http://www.ctu.mrc.ac.uk/our_research/research_areas/tuberculosis/studies/stream_stage2/
- See also: The International Union Against Tuberculosis and Lung Disease web page containing information on the trial — http://www.theunion.org/what-we-do/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were assessed for eligibility from 13 hospital clinics in seven countries, and were randomised between March 2016 and January 2020
Pre-assignment Details: 1436 participants were screened and 588 were randomly assigned to treatment.
Groups:
- Regimen A (Long Regimen): Locally used regimen recommended by WHO in 2011
- Regimen B (Control Regimen): Regimen B is based on the regimen described by Van Deun 2010. With Version 8.0 of the protocol Regimen B (Regimen Bmox) is modified by replacement of moxifloxacin with levofloxacin (Regimen Blev). Regimen B without specification of which fluoroquinolone is in the regimen refers to either (Bmox or Blev).
  Product and dose for [<33 kg, 33-50kg, >50 kg] respectively:
  Moxifloxacin [400mg, 600mg, 800mg] OR Levofloxacin [750mg, 750mg,1000mg]; Clofazimine [50mg,100mg,100mg]; Ethambutol [800mg,800mg,1200mg]; Pyrazinamide [1000mg,1500mg, 2000mg]; Isoniazid 300mg, 400mg, 600mg]; Prothionamide [250mg,500mg,750mg]; Kanamycin [15mg per kilogram body weight (maximum 1g)].
- Regimen C (Oral Regimen): Regimen C is a 40-week all-oral regimen consisting of bedaquiline, clofazimine, ethambutol, levofloxacin, and pyrazinamide given for 40 weeks supplemented by isoniazid and prothionamide for the first 16 weeks (intensive phase).
  Product and dose for [<33kg, 33-50kg, >50 kg] respectively:
  Bedaquiline 400mg once daily for first 14 days/200 mg thrice weekly thereafter; Levofloxacin [750mg, 750mg,1000mg]; Clofazimine [50mg, 100mg, 100mg]; Ethambutol [800mg, 800mg, 1200mg]; Pyrazinamide [1000mg,1500mg, 2000mg]; Isoniazid [300mg, 400mg, 600mg]; Prothionamide [250mg, 500mg,750mg].
- Regimen D (6-month Regimen): Regimen D is a 28-week regimen consisting of bedaquiline, clofazimine, levofloxacin, and pyrazinamide given for 28 weeks supplemented by isoniazid and kanamycin for the first 8 weeks (intensive phase).
  Product and dose for [<33kg, 33 to<40kg, 40-50kg, >50-60 kg, >60 kg] respectively:
  Bedaquiline 400mg once daily for first 14 days/200mg thrice weekly thereafter; Levofloxacin [750mg, 750mg, 750mg, 1000mg, 1000mg]; Clofazimine [50mg, 100mg, 100mg, 100mg, 100mg]; Pyrazinamide [1000mg,1500mg, 1500mg, 2000mg, 2000mg]; Isoniazid [400mg, 500mg, 600mg, 800mg, 900mg]; Kanamycin [15 mg per kilogram body weight (maximum 1g)].
Period: Overall Study
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
Started | 32 | 202 | 211 | 143
Completed | 0 | 187 | 196 | 134
Not Completed | 32 | 15 | 15 | 9
Not completed — Protocol Violation | 3 | 6 | 9 | 4
Not completed — No positive culture/no baseline sample | 3 | 9 | 6 | 5
Not completed — Completed but not analysed as recruitment stopped to this arm | 26 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen) | Total
Number analyzed (Participants) | 32 | 202 | 211 | 143 | 588
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.0 [26.0 to 42.0] | 32.8 [25.7 to 40.6] | 32.8 [26.9 to 42.8] | 30.8 [25.5 to 41.6] | 32.7 [26. to 42.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 81 | 79 | 59 | 236
  Male | 15 | 121 | 132 | 84 | 352
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mongolia | 11 | 46 | 48 | 25 | 130
  South Africa | 6 | 28 | 32 | 26 | 92
  Uganda | 0 | 22 | 25 | 9 | 56
  Moldova | 4 | 25 | 26 | 8 | 63
  Georgia | 0 | 13 | 12 | 7 | 32
  Ethiopia | 6 | 21 | 20 | 20 | 67
  India | 5 | 47 | 48 | 48 | 148

OUTCOME MEASURES:

1. Primary Outcome: STREAM Stage 2 Primary Outcome Measure (the Proportion of Patients With a Favourable Outcome at Week 76)
Description: The primary efficacy outcome of the STREAM Stage 2 comparison is status at Week 76 i.e. the proportion of patients with a favourable outcome at Week 76
Time Frame: 76 weeks
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
Number analyzed (Participants) | 0 | 187 | 196 | 134
Participants | 0 | 133 | 162 | 122

2. Other Pre Specified Outcome: Favourable Outcome After Long-term Follow-up (132 Weeks)
Description: The proportion of patients with a favourable outcome at their last efficacy visit
Time Frame: Last efficacy visit, between 96 and 132 weeks
Population: mITT population, assessable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
Number analyzed (Participants) | 26 | 181 | 190 | 128
Participants | 17 | 126 | 152 | 115

3. Other Pre Specified Outcome: Proportion of Patients With Acquired Drug Resistance
Description: The proportion of patients with acquired drug resistance (any drug)
Time Frame: 132 weeks
Population: mITT population, excluding the long regimen (arm A)
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
Number analyzed (Participants) | 0 | 187 | 196 | 134
Participants | 0 | 5 | 5 | 3

4. Other Pre Specified Outcome: Failure or Recurrence (FoR)
Description: probable or definite failure or recurrence (FoR)
Time Frame: final efficacy week (between 96 and 132 weeks)
Population: mITT population, comparing oral to control regimen
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
Number analyzed (Participants) | 0 | 187 | 196 | 0
Participants | 0 | 17 | 4 | 0
Statistical Analysis 1: Comparison: Regimen B (Control Regimen) vs Regimen C (Oral Regimen); Test type: Superiority; p = 0.0016, Log Rank; Cox Proportional Hazard = 0.20, 95% CI 2-sided [0.07 to 0.61]

5. Other Pre Specified Outcome: Failure or Recurrence (FoR)
Description: The proportion of patients with failure or recurrence (FoR)
Time Frame: 132 weeks, control regimen (arm B) using concurrent controls only
Population: mITT population, control regimen (arm B) using only concurrent controls
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
Number analyzed (Participants) | 0 | 127 | 0 | 134
Participants |  | 14 |  | 2
Statistical Analysis 1: Comparison: Regimen B (Control Regimen) vs Regimen D (6-month Regimen); Control regimen (arm B) uses concurrent controls only; Test type: Superiority; p = 0.0005, Log Rank; Cox Proportional Hazard = 0.11, 95% CI 2-sided [0.03 to 0.50]

ADVERSE EVENTS:
Time Frame: 132 weeks
Description: Adverse events reported include all Grade 3 and 4 events, which may overlap with the reporting of the Serious Adverse Events.
Arm/Group | Regimen A (Long Regimen) | Regimen B (Control Regimen) | Regimen C (Oral Regimen) | Regimen D (6-month Regimen)
All-Cause Mortality (participants affected / at risk) | 0/32 | 8/202 | 11/211 | 2/143
Serious Adverse Events (participants affected / at risk) | 8/32 | 44/202 | 44/211 | 33/143
Other Adverse Events (participants affected / at risk) | 21/32 | 114/202 | 109/211 | 82/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Long Regimen) (N=32) | Regimen B (Control Regimen) (N=202) | Regimen C (Oral Regimen) (N=211) | Regimen D (6-month Regimen) (N=143)
Hearing and vestibular disorders (SMQ) (Ear and labyrinth disorders) | 0 (0) | 7 (7) | 7 (7) | 7 (7)
General disorders and administration site conditions (General disorders) | 1 (1) | 6 (6) | 2 (2) | 6 (6)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 5 (5) | 2 (2)
Investigations (Investigations) | 1 (1) | 3 (3) | 4 (4) | 5 (5)
Hepatic disorders (SMQ) (Hepatobiliary disorders) | 1 (1) | 5 (5) | 4 (4) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Social circumstances (Social circumstances) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Psychiatric disorders (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Torsade de pointes/QT prolongation (SMQ) (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 12 (12) | 9 (9) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Long Regimen) (N=32) | Regimen B (Control Regimen) (N=202) | Regimen C (Oral Regimen) (N=211) | Regimen D (6-month Regimen) (N=143)
Torsade de pointes/QT prolongation (SMQ) (Cardiac disorders) | 2 (2) | 47 (47) | 52 (52) | 38 (38)
Hepatic disorders (SMQ) (Hepatobiliary disorders) | 3 (3) | 31 (31) | 33 (33) | 15 (15)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 10 (10) | 22 (22) | 30 (30) | 20 (20)
Investigations (Investigations) | 10 (10) | 25 (25) | 19 (19) | 14 (14)
Hearing and vestibular disorders (SMQ) (Ear and labyrinth disorders) | 2 (2) | 20 (20) | 9 (9) | 6 (6)
General disorders and administration site conditions (General disorders) | 0 (0) | 5 (5) | 4 (4) | 6 (6)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 3 (3) | 6 (6)
Infections and infestations (Infections and infestations) | 0 (0) | 8 (8) | 3 (3) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 2 (2) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 6 (6)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Psychiatric disorders (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation of the trial is that the open-label design might have influenced decisions on regimen change, especially for non-bacteriological reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT02409290/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02409290/SAP_001.pdf